CLINICAL TRIAL: NCT03889379
Title: Albuterol and Immune Cell Composition
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Team decided not to initiate study.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 181229451
Record Dates: First submitted 2019-01-31; First posted 2019-03-26 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Immune Cell Composition
Keywords: albuterol; immune cells; immune cell composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Effects of Albuterol on Immune Cell Composition (Experimental): This is a single subject repeated measure experimental design with each participant acting as his/her own control.
  Interventions: Drug: Administration of albuterol

INTERVENTIONS:
Drug: Administration of albuterol — Participants will inhale nebulized albuterol at a concentration of 2.5mg diluted in 3mL of normal saline for 20 minutes.

SUMMARY:
The aim of this pilot study is to determine the effects of albuterol on the composition of immune cells in the bloodstream for possible future use in patients with neuroblastoma.

DETAILED DESCRIPTION:
Neuroblastoma is a cancer that typically affects the nerves of children. Sometimes the treatment required for neuroblastoma is an autologous stem cell transplant, where patients who are experiencing neuroblastoma will undergo an expansion of their blood system and collect their peripheral blood to later infuse back into them after chemotherapy and/or radiation. However, up to 14% of individuals experience complications with this procedure.

Research has shown that certain drugs that cause similar effects on the body to that of acute exercise can elicit a more favorable donation. However, these drugs are very costly. Albuterol, on the other hand, is a regularly used drug that may have a similar effect on the body as adrenaline and is used to treat individuals who are experiencing respiratory airway distress. The benefit of albuterol is that it can be administered through inhalation, further reducing patient burden.

The aim of this pilot study is to determine the effects of albuterol on the composition of immune cells in the bloodstream. Five healthy volunteers (age 21-44 years) will be recruited to participate in this study. Each participant will donate a 6ml blood sample before and during a 20-minute continuous albuterol nebulization through an IV catheter. During the last 10 minutes of the nebulization, participants will submit to another 6mL blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* 21-44 years of age

Exclusion Criteria:

* Subjects must not: be younger than 21 or older than 44 years of age
* Indicate a condition on the ACSM-AHA preexercise screening questionnaire indicating that physician approval is required prior to exercise
* current user of tobacco products or have quit within the previous 6-months
* body mass index of >30 kg/m2, or waist girth of >102cm for men and >88cm for women
* use over-the-counter medication known to affect the immune system (i.e. regular use of ibuprofen/aspirin, anti-histamines or beta-blockers)
* have chronic/debilitating arthritis
* have been bedridden in the past three months
* have common illness (i.e. colds) within the past 6-weeks
* have HIV
* have hepatitis
* have had a stroke
* have major affective disorder
* have any autoimmune disease
* have central or peripheral nervous disorders
* have blood vessel disease
* have cardiovascular disease (CVD)
* use of any prescription medication
* pregnancy or are breast-feeding
* asthma, emphysema, bronchitis, kidney disease; pheochromocytoma; diabetes; overactive thyroid
* history of severe anaphylactic reaction to an allergen
* or are scheduled to have surgery
* Individuals who pass the exclusion criteria detailed above but present with more than one of the following CVD risk factors will also be excluded from the study: family history of myocardial infarction, coronary revascularization, or sudden death before 55 years of age in father or other male first-degree relative or before 65 years of age in mother or other female first-degree relative; hypertension (systolic blood pressure of >140 mmHg or diastolic blood pressure >90 mmHg); dyslipidemia (total serum cholesterol of >200 mg/dl); pre-diabetes (fasting blood glucose of >100mg/dl but <126 mg/dl).

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
Quantification of NK Cells (CD3-/CD56+). | One year
  Investigators will collect a 6mL blood sample into EDTA anti-coagulant tubes before and during the last five minutes of an albuterol nebulization to assess the quantification in both absolute number and proportion of NK cells (CD3-/CD56+) using a MACSQuant flow cytometer and subsequent analysis on FlowLogic Software (v7.2.1). The last five minutes of nebulization of blood sample will be directly compared to the pre nebulization blood sample in the same participants in the same research arm.
Quantification of Gamma Delta T Cells (CD4-CD8-). | One year
  Investigators will collect a 6mL blood sample into EDTA anti-coagulant tubes before and during the last five minutes of an albuterol nebulization to assess the quantification in both absolute number and proportion of Gamma Delta T cells (CD3+/CD4-/CD8-) using a MACSQuant flow cytometer and subsequent analysis on FlowLogic Software (v7.2.1). The last five minutes of nebulization of blood sample will be directly compared to the pre nebulization blood sample in the same participants in the same research arm.
Quantification of Gamma T cell subsets (CD3+/CD4/CD8). | One year
  Investigators will collect a 6mL blood sample into EDTA anti-coagulant tubes before and during the last five minutes of an albuterol nebulization to assess the quantification in both absolute number and proportion of T-cell subsets (CD3+/CD4/CD8) using a MACSQuant flow cytometer and subsequent analysis on FlowLogic Software (v7.2.1). The last five minutes of nebulization of blood sample will be directly compared to the pre nebulization blood sample in the same participants in the same research arm.

CONTACTS AND LOCATIONS:
Overall Officials: Grace M Niemiro, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided